CLINICAL TRIAL: NCT00646438
Title: United States CABG Diabetes Project (USCDP) Pilot Study
Brief Title: United States Coronary Artery Bypass Surgery (CABG) Diabetes Project (USCDP) Pilot Study
Acronym: USCDP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Providence Heart & Vascular Institute (Other)
Collaborators: Sanofi (Industry); LifeScan (Industry)
Responsible Party: Anthony Furnary, MD / Principal Investigator, Providence Heart & Vascular Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: USCDP
Record Dates: First submitted 2008-03-25; First posted 2008-03-28 (Estimated); Last update posted 2009-02-04 (Estimated); Status verified 2008-03

CONDITIONS: Diabetes; Coronary Artery Disease
Keywords: Diabetes; CABG
MeSH Terms: conditions — Diabetes Mellitus; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): strict glucose control (study arm)
  Interventions: Drug: Strict Glycemic Control for one year post-op CABG
- 2 (No Intervention): standard insulin treatment (control arm)

INTERVENTIONS:
Drug: Strict Glycemic Control for one year post-op CABG — The CDE and Study Coordinator will also meet with the patient in the hospital to show how the Lifescan One-Touch Ultra II glucometer works and review the study follow-up schedule. Patients will be sent home with the Lifescan One-Touch Ultra II glucometer and a supply of strips.
  Post-Discharge Period Patients will meet alternatively with the CDE and study doctor on a specific schedule including every week for the first month, every 2 weeks in the second month, and every month thereafter till the 12th month. During these sessions the BG records will be downloaded from the Lifescan One-Touch Ultra II glucometer and reviewed to see patterns and any areas that could be improved or changed.
  For all patients in the study arm, the medications that are being taken and the results of glucose monitoring charts will be reviewed weekly with endocrinologists so that any additional recommendations may be made to improve glucose control.
  Other Names: USCDP; Portlan Protocol
  Arms: 1

SUMMARY:
Standard care for patients with diabetes having CABG surgery at Providence St. Vincent Medical Center includes strict control of blood sugar (glucose) levels for 3 days after surgery. This is done through frequent monitoring of blood sugar levels and by giving insulin continuously through a needle into a vein (intravenously). This intensive glucose control has resulted in fewer complications such as serious infections and death, and has shortened the length of the hospital stay for patients.

This study treatment is different from standard treatment in that it extends the intensive glucose control beyond the third postoperative day to one full year. Once discharged from the hospital following the CABG procedure, the intense glucose control is done using subcutaneous insulin (a shot under the skin), oral medications, and by measuring blood sugar levels frequently.

The purpose of this study is to see how safe and effective strict glucose control is when extended beyond 3 days and hospital discharge for one year. Another purpose is to see how well patients can comply with the daily management of intensive glucose control for one-year as well as the study follow-up schedule.

DETAILED DESCRIPTION:
Purpose Pilot study to gather information for "United States CABG Diabetes Project" (USCDP) Multi-center Randomized Trial.

For 14 years our research team has successfully implemented an increasingly aggressive series of intravenous insulin protocols that normalize blood glucose levels for 3 postoperative days in patients with diabetes who undergo cardiac surgery. This has resulted in significant reductions in mortality, infection and length of stay (LOS) and has normalized those outcomes to those of the population without diabetes (DM). The current protocol ends on the morning of the 3rd postoperative day.

We believe that a logical expansion of this groundbreaking work is to extend the duration of intensive glycemic control beyond the third postoperative day and into the outpatient period. However it would be impossible to do so with the continued use of CII therapy. Therefore, we propose to employ intensive subcutaneous insulin therapies and oral hypoglycemic agents to affect continued tight glycemic control following discontinuation of CII and continue such therapy beyond hospital discharge for a period of at least one year.

We hypothesize that this will lead to further reductions in major adverse cardiac outcomes in the high-risk diabetes coronary artery bypass grafts (CABG) subgroup. The optimal method to test this hypothesis is with a very large, multi-center clinical trial. However, before embarking on such a resource-consuming endeavor, we intend to test the concepts, methods, implementation strategies, patient acceptability and compliance, proposed biomarkers and clinical outcomes of such a trial with this proposed limited pilot study.

If the information obtained from this pilot study is favorable, we will submit for full funding of the multicenter USCDP clinical trial to the NIDDK and NHLBI divisions of the NIH. In order to test all aspects of the proposed trial, we intend to randomize patients into this pilot study.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 - 80 years old
* Pre-op diagnosis of diabetes
* Scheduled for elective or urgent CABG surgery
* Able to sign informed consent for research study

Exclusion Criteria:

* Patients less than 18 years old or greater than 80 years old
* Emergent or salvage CABG surgery
* Other surgical intervention planned in same setting ( Valve surgery, TMR, MAZE...)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2009-03; Primary Completion 2012-02 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
The purpose of this study is to see how safe and effective strict glucose control is when extended beyond 3 days and hospital discharge for one year. | 3 years

SECONDARY OUTCOMES:
Another purpose is to see how well patients can comply with the daily management of intensive glucose control for one-year as well as the study follow-up schedule. | 3 Years

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Furnary, MD, Principal Investigator — Providence Heart & Vascular Institute
Locations (1):
- Providence St. Vincent Medical Center, Portland, Oregon, United States